CLINICAL TRIAL: NCT01682902
Title: A Randomised Trial Evaluating Continuous Subcutaneous Infusion of Formulations of NN1218 and NovoLog® in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3930; U1111-1121-5106 (Other: WHO)
Record Dates: First submitted 2012-08-31; First posted 2012-09-11 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation 1 (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Formulation 2 (Experimental)
  Interventions: Drug: Faster-acting insulin aspart
- Insulin aspart (NovoLog®) (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Administration: Subcutaneous infusion. The subjects will remain on their own pump during the trial. Subjects will have blinded continuous glucose monitoring (CGM) throughout the trial (3 treatment periods of 14 days) and meal tests consisting of a standardised breakfast (liquid meal) will be performed on the 14th day of each treatment period.
  Other Names: NN1218
  Arms: Formulation 1
Drug: Faster-acting insulin aspart — Administration: Subcutaneous infusion. The subjects will remain on their own pump during the trial. Subjects will have blinded continuous glucose monitoring (CGM) throughout the trial (3 treatment periods of 14 days) and meal tests consisting of a standardised breakfast (liquid meal) will be performed on the 14th day of each treatment period.
  Other Names: NN1218
  Arms: Formulation 2
Drug: insulin aspart — Administration: Subcutaneous infusion. The subjects will remain on their own pump during the trial. Subjects will have blinded continuous glucose monitoring (CGM) throughout the trial (3 treatment periods of 14 days) and meal tests consisting of a standardised breakfast (liquid meal) will be performed on the 14th day of each treatment period.
  Arms: Insulin aspart (NovoLog®)

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to evaluate continuous subcutaneous infusion of NN1218 formulations and NovoLog® in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (diagnosed clinically) for at least 12 months prior to the screening visit (Visit 1)
* Treatment with the same insulin analogue by CSII (continuous subcutaneous insulin infusion) for the previous 3 months prior to the screening visit (Visit 1)
* Using a MiniMed Paradigm® pump (515/715, 522/722 or 523/723) for the previous 6 months prior to the screening visit (Visit 1)
* Glycosylated haemoglobin (HbA1c) below or equal to 9.0% by central laboratory
* Body Mass Index (BMI) below or equal to 35.0 kg/m^2

Exclusion Criteria:

* History of diabetic ketoacidsosis (DKA) episodes requiring hospitalization within 6 months prior to the screening visit (Visit 1)
* History of abscess at the infusion site within 6 months prior to the screening visit (Visit 1)
* Hypoglycaemic unawareness as judged by the Investigator or history of severe hypoglycaemic episodes requiring hospitalization within the last 6 months prior to the screening visit (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mean change in plasma glucose concentration | From 0-2 hours after administration of standardised meal after the first, the second, and the third 14-day treatment period

SECONDARY OUTCOMES:
Self-measured plasma glucose (SMPG) 7-point profile | After the first, the second, and the third 14-day treatment period
Self-measured plasma glucose (SMPG) 9-point profile | After the first, the second, and the third 14-day treatment period
Number of adverse events (AEs) (including infusion site reactions/infections) | Days 0-14 for each treatment periods
Number of hypoglycaemic episodes | Days 0-14 for each treatment period
Number of unexplained self-reported episodes of hypoglycaemia or hyperglycaemia (confirmed by SMPG) | Days 0-14 for each treatment period
Number of episodes of infusion set occlusions | Days 0-14 for each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Atlanta, Georgia, United States

REFERENCES:
- [Result] Bode BW, Johnson JA, Hyveled L, Tamer SC, Demissie M. Improved Postprandial Glycemic Control with Faster-Acting Insulin Aspart in Patients with Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion. Diabetes Technol Ther. 2017 Jan;19(1):25-33. doi: 10.1089/dia.2016.0350. Epub 2017 Jan 5. PMID 28055230
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com